CLINICAL TRIAL: NCT04771208
Title: I Kua na'u "Let Me Carry Out Your Last Wishes" Advance Care Planning for Native Hawaiian Elders - Trial Phase
Brief Title: I Kua na'u Advance Care Planning for Native Hawaiian Elders
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); University of Hawaii (Other); Queen's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-41343; 1R01NR018400 (NIH)
Record Dates: First submitted 2021-02-20; First posted 2021-02-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Advance Care Planning
Keywords: medical decision making; Native Hawaiians; educational decision aid video; doctor patient communication

STUDY DESIGN:
Intervention Model Description: There are 2 different study designs included:
  1. Pre-post study: NH participants from Homestead and Group Assisted Living (N=110) will partake in a pre-post study design. Participants will receive a baseline survey (as described below), view the ACP video intervention, and receive a post-intervention survey, which includes the same items as the baseline survey.
  2. RCT: In the ambulatory clinics we will conduct a randomized controlled trial (N=110), and randomize (1:1) in blocks of 2 and 4 to either the video (intervention) or usual care (control) arm. The intervention group will use the ACP video decision aid and participants in the control group will receive usual care. All participants will have a baseline survey, be randomized to intervention or control, and receive a post-intervention survey, which includes the same items as the baseline survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pre-Post Trial (Other): Native Hawaiian participants from Homestead and Group Assisted Living (N=110) will partake in a pre-post study design. Participants will receive a baseline survey (as described below), view the ACP video intervention, and receive a post-intervention survey, which includes the same items as the baseline survey. In-person or phone interviews will be done at three and six months.
  Interventions: Behavioral: I kua na'u "Let Me Carry Out Your Last Wishes"
- Randomized Clinical Trial: Control Group (No Intervention): In the ambulatory clinics we will conduct a randomized controlled trial (N=110), and randomize (1:1) to either the video (intervention) or usual care (control) arm. The control group will receive usual care. All participants will have a baseline survey, be randomized to intervention or control, and receive a post-intervention survey, which includes the same items as the baseline survey. Follow-up in person or by phone interviews will be done at three and six months.
- Randomized Clinical Trial: Intervention Group (Experimental): In the ambulatory clinics we will conduct a randomized controlled trial (N=110), and randomize (1:1) to either the video (intervention) or usual care (control) arm. The intervention group will use the ACP video decision aid. All participants will have a baseline survey, be randomized to intervention or control, and receive a post-intervention survey, which includes the same items as the baseline survey. Follow-up in person or by phone interviews will be done at three and six months.
  Interventions: Behavioral: I kua na'u "Let Me Carry Out Your Last Wishes"

INTERVENTIONS:
Behavioral: I kua na'u "Let Me Carry Out Your Last Wishes" — A combination of Native Hawaiian advance care planning video decision support tool and personalized video declarations shared with providers and family members.
  Arms: Pre-Post Trial; Randomized Clinical Trial: Intervention Group

SUMMARY:
Communication surrounding serious illness decision making is formalized in Advance Care Planning (ACP), a process involving verbal or written information designed to inform patients of possible medical options including palliative and hospice care services. Numerous studies have suggested that improved ACP rates better align health care delivery with patient preferences. Despite expansion of ACP services in the health care system, Native Hawaiians (NHs) consistently have negligible rates of ACP and low use of palliative and hospice care services. To address these shortcomings, our multi-disciplinary community and research group has partnered to create the I kua na'u "Let Me Carry Out Your Last Wishes" ACP video intervention. Our Community-Based Collaborative Approach will create, develop and test the I kua na'u comprehensive video-based ACP program honoring the history, opinions, and culture of NHs. Indeed, NH culture is primarily an oral tradition in which the spoken word permeates the life of NHs and is the normal way of interacting with neighbors, including in its most recent adaptation with the use of video media. The I kua na'u program will include videos tailored for the different settings in which older NHs live and get medical care. The videos will explain the importance of ACP, empower NHs to tell their story ('olelo Kama'ilio; "Talk Story") by allowing the recording of personal video declarations of ACP wishes, and the ability to share the personal video declaration with family, friends and clinicians. The overall objective is to conduct a five-year program that includes two years of development of the I kua na'u ACP video program with focus group testing, and then three years of implementation in the NH community. Demonstrating the effectiveness of using the video program in NHs represents an essential step to implement this tool in practice. The Specific Aim is to compare the ACP engagement, knowledge, decisional conflict, and ACP completion rates in 220 NHs over the age of 55 in: (a) a pre-post study design in 110 people living on Homestead or Assisted Living using the video intervention, and (b) a randomized trial of 110 people recruited from Ambulatory Clinics.

DETAILED DESCRIPTION:
This project entitled, "I kua na'u" in Hawaiian, translates to "Let me carry out your last wishes." This work aims to honor the Native Hawaiian (NH) sense of cultural context for initiating a conversation between elders and their families through a video intervention to promote Advance Care Planning (ACP) in a manner that respectfully communicates the personal preferences of NH elders to their family, caregivers and the health care system. The full I kua na'u program will examine a video enhanced intervention designed by and for Native Hawaiians (NH) and their family caregivers in three distinct settings: 1) NH Homesteads, 2) Assisted Living, and 3) Ambulatory Clinics. The overall objective of the present proposal is to conduct the first phase of the program, which covers the planned two year development period of the I kua na'u ACP video program. During this time, we will conduct a series of focus groups and one-on-one stakeholder interviews to inform the creation of: A) NH ACP videos; B) a NH personal video declaration process; and, C) NH community members training program to deliver the intervention.

Native Hawaiians (NHs), the indigenous people of Hawai'i, comprise a diverse population of more than 500,000 individuals living in the US and are one of the fastest growing racial/ethnic groups in the country. The highest concentration (55%) of NHs live in the State of Hawai'i, the ancestral home of all NH people. Several studies have established a higher mortality rate among NHs that occurs at an age 10-15 years earlier than the general US population. A recent study found that NHs had the lowest life expectancy of the five major ethnic groups in the state of Hawai'i, with a consistent 10-year gap between NHs and the longest living ethnic group. According to the US Census 2010, ~100,000 NHs over the age of 50 currently live in the US with 60% residing in the State of Hawai'i. Yet few studies have examined the use of end-of-life care and advance care planning in NHs who are at high risk for more frequent and earlier age death. Thus, this proposal aims to fill the gap in our understanding of ACP among NH elders and will develop, test and disseminate a culturally informed intervention to improve ACP practices among NH elders and their families.

Mounting evidence suggests that NHs rarely participate in ACP or communicate their ACP wishes to their families, who are often the primary caregivers. Palliative care and hospice services have been associated with less intensive interventions at the end of life, possibly due to improved communication and decision making. Learning about ACP and communicating with family and providers is the best way for a person to get health care that is concordant with one's wishes and values. NHs represent a unique population with distinct cultural, epidemiological, genetic, and psychosocial characteristics. Evidence suggests that they also have distinct health care and health communication preferences. Although some of these distinct features and preferences may contribute to disparities in health care for NHs with advanced illness, these disparities may also be due to identified health communication gaps.

While the topic of ACP communication specifically is understudied, critical health communication gaps exist for many NHs. Previous research by members of this study team and others have identified relevant health communication challenges in NH communities. For instance, practical challenges included jargon and lack of plain English. Interpersonal issues included doctors rushing, doctors not assessing comprehension, and doctors not treating respondents as people. Respondents noted that they would often not ask questions even when they knew they did not understand because they did not want the provider to think negatively of them. Overarching themes to improve communication gaps included: the importance of family and community in health information dissemination, the importance of personal experience and relationships to the salience of health information, and the desire for local cultural relevance in health communication.

ACP seeks to ensure that patients receive medical care consistent with their values, goals and preferences during the advanced stages of a disease when they no longer have capacity to make decisions. ACP is the most consistent factor associated with better end-of-life outcomes in patients with advanced illness and their caregivers. The lack of ACP is associated with more aggressive interventions, more terminal hospitalizations, lower hospice use, and worse caregiver burden and family bereavement outcomes. Unfortunately, ACP completion remains inadequate, and has remained consistently low. Studies show that traditional written and verbal ACP does not effectively inform many patients and caregivers, and often occurs late in the disease process, which is especially true in vulnerable communities such as NHs. Other common barriers to ACP include lack of tailoring for NHs, variable quality of clinician communication, complex relationships between families and clinicians regarding decision making, and the inability for patients to realistically envision accurate future health states. These barriers present challenges as well as an opportunity. This opportunity for change is a major goal of this proposal to evaluate not just an intervention and its meaningfulness to individuals, caretakers, and family, but also, to educate and train our communities on how to deploy the intervention in real world settings. Individuals from our NH communities will be trained to carry out the intervention and to implement this training using our community peer-to-peer model.

ELIGIBILITY:
Subject Inclusion criteria:

1. NH adult > 55 years of age;
2. Pre-existing relationship with a primary care provider (PCP, minimum of two prior visits to PCP);
3. Referral by collaborating community organization.

Subject Exclusion Criteria:

1. inability to view videos due to visual impairment (worse than 20/200 corrected);
2. psychological state not appropriate for ACP discussions as determined by RA or clinician;
3. cognitive impairment (≥2 errors) as assessed by the validated Short Portable Mental Status Questionnaire.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in ACP Knowledge (Pre-Post Trial) | Baseline, 6 weeks, 3 months, 6 months
  Six questions regarding knowledge of ACP which were used and validated in previous studies will be asked. A score of 0-6 will be assigned. Higher scores indicate more knowledge. Questions will be asked before and after the intervention is administered.
Change in ACP Knowledge (RCT) | Baseline, 6 weeks, 3 months, 6 months
  Six questions regarding knowledge of ACP which were used and validated in previous studies will be asked. A score of 0-6 will be assigned. Higher scores indicate more knowledge.

SECONDARY OUTCOMES:
Change in End of Life Health Care Preferences (Pre-Post Trial) | Baseline, 6 weeks, 3 months, 6 months
  Participants will be asked 2 questions about their end of life health care preferences. Any change in response will be coded as a change. Questions will be asked before and after the intervention is administered.
Change in Decisional Conflict (Pre-Post Trial) | Baseline, 6 weeks, 3 months, 6 months
  Decisional conflict will be measured with a 2 question survey that returns a score of 0-10. Higher scores indicate more conflict. Questions will be asked before and after the intervention is administered.
Change in Advance Care Planning Engagement (Pre-Post Trial) | Baseline, 6 weeks, 3 months, 6 months
  Four validated likert scale questions regarding ACP engagement are averaged to return an overall score of 0-5. Higher scores indicate increased engagement. Questions will be asked before and after the intervention is administered.
Change in End of Life Health Care Preferences (RCT) | Baseline, 6 weeks, 3 months, 6 months
  Participants will be asked 2 questions about their end of life health care preferences. Any change in response will be coded as a change. Comparison will be post-intervention vs control.
Change in Decisional Conflict (RCT) | Baseline, six weeks, 3 months, 6 months
  Decisional conflict will be measured with a 2 question survey that returns a score of 0-10. Higher scores indicate more conflict. Comparison will be post-intervention vs control.
Change in Advance Care Planning Engagement (RCT) | Baseline, six weeks, 3 months, 6 months
  Four validated likert scale questions regarding ACP engagement are averaged to return an overall score of 0-5. Higher scores indicate increased engagement. Comparison will be post-intervention vs control.
Consumer Assessment of Healthcare Providers and Systems Survey (RCT) | 6 weeks post enrollment
  11 questions from the validated AHRQ survey that asks patients to report on their experiences with providers and staff in primary care settings.
Consumer Assessment of Healthcare Providers and Systems Survey (Pre-Post Trial) | 6 weeks post enrollment
  11 questions from the validated AHRQ survey that asks patients to report on their experiences with providers and staff in primary care settings.
Video Preferences (RCT) | 6 weeks post enrollment
  4 questions to determine the participant's level of comfort in watching the video.
Video Preferences (Pre-Post Trial) | 6 weeks post enrollment
  4 questions to determine the participant's level of comfort in watching the video.
ACP Documentation (RCT) | 12 months post enrollment
  2 questions about whether the participant has had a conversation about ACP with either a provider or a friend/family member, as well as a EHR review for specific documentation of ACP preferences (intubation, DNR, dialysis, POLST, health care proxy).
ACP Documentation (Pre-Post Trial) | 12 months post enrollment.
  2 questions about whether the participant has had a conversation about ACP with either a provider or a friend/family member.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Paasche-Orlow, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- University of Hawaii, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quintiliani LM, Kamaka M, Henault L, Antonio MCK, Sentell T, Spencer K, Akaka G, Honda LKL, Hanakeawe D, Dillard A, Kekauoha BP, Davis AD, Seitz R, Cabral HJ, Volandes A, Leimomi Mala Mau MK, Paasche-Orlow MK. I kua na'u "Let me carry out your last wishes" Clinical trial protocol to promote advance care planning among native Hawaiian populations. Contemp Clin Trials. 2023 Dec;135:107365. doi: 10.1016/j.cct.2023.107365. Epub 2023 Oct 24. PMID 37884121